CLINICAL TRIAL: NCT02513407
Title: Reducing Cancer and Chronic Disease Risk in Medically Vulnerable Communities: A Feasibility Study Measuring Behavioral and Biological Outcomes of the Eat Move Live Intervention
Brief Title: Eat, Move, Live Intervention in Reducing Chronic Disease Risk in Medically Vulnerable Communities
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 15160; NCI-2015-01220 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 15160 (Other: City of Hope Medical Center)
Record Dates: First submitted 2015-07-29; First posted 2015-07-31 (Estimated); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Healthy Subject
MeSH Terms: interventions — Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group I (EML) (Experimental): Participants complete an assessment on knowledge, attitudes, and behaviors at baseline and attend 2 weekday sessions comprised of interactive education segment that is culturally responsive, and based on the community EML program, and topics including: nutrition guideline, nutrition label reading, comparison shopping/grocery store tour, recipe modification and healthy food preparation, eating healthy on a budget, and making healthy choices outside the home (e.g., restaurants) and physical activity over 1 hour led by CHE, a physical activity conducted by Duarte Fitness Centers instructors over 30 minutes, and cooking/taste test demonstration co-led by the CHE and local chef over 30 minutes over 12 weeks. Participants are also prescribed and encouraged to participate in 3 days a week exercise classes (for > 30 minutes) including salsa, Zumba and other aerobic exercises that are provided at Duarte Fitness Center.
  Interventions: Behavioral: Behavioral Dietary Intervention; Other: Educational Intervention; Behavioral: Exercise Intervention; Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration
- Group II (control) (Active Comparator): Participants receive a fitness tracker to track their physical activity and be wait listed to receive the intervention during month 10-12.
  Interventions: Behavioral: Behavioral Dietary Intervention; Behavioral: Exercise Intervention; Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration

INTERVENTIONS:
Behavioral: Behavioral Dietary Intervention — Attend healthy nutritional education session
Other: Educational Intervention — Attend EML educational session
  Other Names: Education for Intervention; Intervention, Educational
  Arms: Group I (EML)
Behavioral: Exercise Intervention — Attend exercise educational session
  Arms: Group I (EML)
Behavioral: Exercise Intervention — Receive fitness tracker
  Arms: Group II (control)
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized pilot research trial studies how well Eat, Move, Live (EML) works in reducing chronic disease risk in medically vulnerable communities. Obesity, unhealthy diet, and physical inactivity are linked to increased cancer risk, especially hormone-related cancer (example, breast cancer). Improving healthy lifestyle practices, namely increasing physical activity and encouraging healthy eating behaviors may reduce the risk of getting cancer and chronic disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Level of exercise.

II. Reduction in barriers to exercise.

III. Level of self-reported 5-9 servings of fruits and vegetables consumption.

IV. Reduction in barriers to fruit and vegetable consumption.

V. Improvement in biologic/metabolic markers such as hemoglobin A1c, fasting plasma glucose, and body weight.

OUTLINE: Participants are randomized to 1 of 2 groups.

GROUP I: Participants complete an assessment on knowledge, attitudes, and behaviors at baseline and attend 2 weekday sessions comprised of interactive education segment that is culturally responsive, and based on the community EML program, and topics including: nutrition guideline, nutrition label reading, comparison shopping/grocery store tour, recipe modification and healthy food preparation, eating healthy on a budget, and making healthy choices outside the home (e.g., restaurants) and physical activity over 1 hour led by Certified Health Educator (CHE), a physical activity conducted by Duarte Fitness Centers instructors over 30 minutes, and cooking/taste test demonstration co-led by the CHE and local chef over 30 minutes over 12 weeks. Participants are also prescribed and encouraged to participate in 3 days a week exercise classes (for > 30 minutes) including salsa, Zumba and other aerobic exercises that are provided at Duarte Fitness Center.

GROUP II: Participants receive a fitness tracker to track their physical activity and be wait listed to receive the intervention during month 10-12.

After completion of study, participants are followed up immediately and at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Mothers/female guardians of elementary aged students
* Self identify as Latina
* Not adherent to the standard for > five servings of fruits and vegetable and 150 minutes of physical activity

Exclusion Criteria:

* Not a parent of elementary aged student in Duarte Unified School District (DUSD)
* Does not self-identify as Latina
* Does not speak/read/write/understand English/Spanish - Diagnosed with diabetes
* Consumes 5+ servings of fruits and vegetables and is active for at least 30 minutes 5+ days per week
* Has a condition or psychological difficulties that affects day-to-day activities
* Has physical limitations and cannot participate in physical activity

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-04-06 (Actual); Primary Completion 2016-10-15 (Actual); Study Completion 2026-08-10 (Estimated)

PRIMARY OUTCOMES:
Changes in plasma glucose level measured using point of care glucometer OneTouch Ultra® 2 | Baseline to up to 3 months
  Will convert plasma glucose into binary outcome variables and evaluate the effect on intervention on these outcomes controlled for significant confounders (age, income, and education will be evaluated for confounding in the logistic regression model). Chi-square goodness of fit tests will compare percent reduction in weight between the control and intervention groups. Chi square tests will be used to determine whether participants reduced weight by 3%. Repeated ANCOVA will be used. Outcome variables will be dichotomized to fit a logistic regression modeling procedures.
Changes in hemoglobin A1c level measured using a point of care device A1CNow® | Baseline to up to 3 months
  Will convert hemoglobin A1c into binary outcome variables and evaluate the effect on intervention on these outcomes controlled for significant confounders (age, income, and education will be evaluated for confounding in the logistic regression model). Chi-square goodness of fit tests will compare percent reduction in weight between the control and intervention groups. Chi square tests will be used to determine whether participants reduced weight by 3%. Repeated ANCOVA will be used. Outcome variables will be dichotomized to fit a logistic regression modeling procedures.
Changes in level of self reported 5-9 servings of fruits and vegetables using self evaluation and the daily food diary | Baseline to up to 3 months
  Chi-square test and Logistic regression analysis will be used to determine whether the intervention significantly motivated participants to consume 7-8 servings of fruits/vegetables per day, adjusting for significant confounders (e.g., age, baseline BMI). Additionally, the Cochran Q test will be used to evaluate changes on barriers to fruit/vegetable consumption at the baseline and follow-up time points.
Changes in reduction in barriers to exercise using self-report evaluation based on historical EML program using Likert-type scale items | Baseline to up to 3 months
  Compliance to exercise at baseline and follow-up will be assessed using Logistic regression analysis. Additionally, the Cochran Q test will be used to evaluate changes on barriers to exercise at the baseline and follow-up time points.
Changes in self-reports of activity tracker readings | Up to 3 months
  Will compare baseline and follow-up exercise levels between the intervention and control groups in an independent t-tests, and compare the pre- to post-intervention change in activity tracker readings between groups with repeated measure analysis of covariance with age and baseline body mass index (BMI) as confounders.
Reduction in barriers to fruit and vegetable consumption using self-evaluation based on historical EML program using Likert-type scale | Baseline to up to 3 months
  Cochran Q test will be used to assess participants' barriers to fruit and vegetable consumption at different follow up period.

CONTACTS AND LOCATIONS:
Overall Officials: Kimlin Ashing-Giwa, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States